CLINICAL TRIAL: NCT06906250
Title: European Venous Registry
Acronym: EVeR
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Baccellieri Domenico, Prof., M.D, IRCCS San Raffaele
Other Study IDs: EVeR- European Venous Registry
Record Dates: First submitted 2025-03-19; First posted 2025-04-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Deep Venous Disease of the Lower Limbs
Keywords: acute or chronic lower limb deep venous disease; iliac and/or common femoral veins; inferior vena cava

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- all patients suffering from deep venous disease of the lower limbs

SUMMARY:
The European Venous Registry (EVeR) is an international repository of data on the treatments and outcomes of people with deep venous disease. The registry is designed to evaluate the outcomes of venous interventions over a ten-year period, with the ultimate goal to inform clinical decision making through the delivery of scientific evidence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an imaging-confirmed new diagnosis of acute or chronic lower limb deep venous disease involving the iliac and/or common femoral veins, with or without extension to the inferior vena cava, or patients with an imaging-confirmed new diagnosis involving the IVC only.
* Consent to enter registry.

Exclusion Criteria:

* Unable to consent to enter into registry.
* Isolated upper limb DVT.
* Central venous thrombosis (e.g. superior vena cava obstruction).
* Isolated deep vein thrombosis below the common femoral vein.
* Isolated superficial venous thrombosis.
* Isolated superficial venous thrombophlebitis.
* Isolated varicose veins.
* Aged <18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population sampled for data collection includes all patients suffering from deep venous disease of the lower limbs who are treated in the centres joining the registry. These include patients receiving surgery as well as those not receiving surgery. Only prospective patients will be allowed.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-05 (Actual); Primary Completion 2034-09-30 (Estimated); Study Completion 2034-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Severity Scores | end of the procedure
  Difference of Clinical efficacy will be evaluated using the Villalta score (range 0-33). The patient was diagnosed as having Post-thrombotic syndrome if the Villalta score was ≥5 or if a venous ulcer was present. A score of 5-9 signifies mild disease, 10-14 moderate disease, and ≥15 severe disease.

SECONDARY OUTCOMES:
Venous Insufficiency Epidemiological and Economic Study/Quality of Life (VEINES-QOL) | 10 years
  Improvement of quality of life will be evaluated using the Veines - qol score.The VEINES-QOL questionnaire consists of 26 items. Each question is standardised using the mean and standard deviation of the sample being coded to give a z-score, these are averaged, and the result transformed to T-scores (mean = 50; standard deviation = 10). High values indicate better outcomes.

CONTACTS AND LOCATIONS:
Locations (10):
- Department of Vascular Surgery, Marseille, France, France
- European Venous Center, Aachen, Germany, Germany
- Clinic of Vascular and Endovascular Surgery at Athens Medical Group, Athens, Greece, Greece
- Interventional Radiology, Galway University Hospitals, Galway, Ireland, Ireland
- IRCCS San Raffaele Hospital, Milan, Italy, Italy
- Department of Vascular and Endovascular Surgery, Erasmus Medical Centre, Rotterdam, Netherlands, Netherlands
- Vascular and Endovascular Department, Viamed Hospitals, Madrid, Spain, Spain
- Department of Cardiovascular Surgery, Acibadem University School of Medicine,, Istanbul, Turkey, Turkey (Türkiye)
- United Kingdom (2):
  - North Bristol NHS Trust, Bristol, United Kingdom
  - St Thomas' Hospital, London, United Kingdom

REFERENCES:
- See also: Related Info — https://esvs.org/ever-venous-registry/